CLINICAL TRIAL: NCT02278146
Title: A Multi-center, Open-label, Prospective, Feasibility Study Evaluating the ParaPatch System for the Treatment of Urinary Incontinence and Overactive Bladder
Brief Title: Feasibility Study Evaluating the ParaPatch System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ParaPatch, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PP-01-2014
Record Dates: First submitted 2014-10-21; First posted 2014-10-29 (Estimated); Results first posted 2017-01-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) Stress urinary incontinence (Experimental): Stress urinary incontinence. Diagnosed with urinary stress incontinence and treated with the ParaPatch System
  Interventions: Device: ParaPatch
- 2) Overactive bladder (Experimental): Overactive bladder. Diagnosed with overactive bladder syndrome and treated with the ParaPatch System
  Interventions: Device: ParaPatch

INTERVENTIONS:
Device: ParaPatch — A device for the treatment of urinary incontinence

SUMMARY:
A multi-center, open-label, prospective, feasibility study evaluating the ParaPatch System for the treatment of urinary incontinence and overactive bladder.

DETAILED DESCRIPTION:
* Baseline Period

  o The baseline period will allow for washout of any medication affecting bladder function and to allow subject to begin her voiding diary.
* Prospective data collection will take place in the form voiding diary. Leak frequency, and other relevant parameters will be collected.
* Inclusion/exclusion criteria will be rechecked at end of baseline.
* Qol questionnaires will be completed in the office at the end of baseline period.
* Evaluation Period

  o During the evaluation period, the subjects will use the ParaPatch System.
* No medications affecting bladder function will be allowed during the evaluation period.
* Subjects will complete voiding diaries, during the evaluation period. Data capture to include: adverse events, medication use, leak frequency and other relevant parameters.
* Qol questionnaires will be completed in the office at the end of evaluation period.
* Follow-up Period

  o Subjects will be followed for after the evaluation period to check for residual Adverse Events.
* No medications affecting bladder function will be allowed during the follow-up period.
* Subjects will be called by the clinical coordinator at the end of the Follow-up period and asked about potential Adverse Events.

ELIGIBILITY:
Inclusion Criteria:

* Women aged from >18 to < 75 years old.
* Subject has the ability to read and comprehend English, and to reliably record information as required by the Protocol, including the proper completion of the questionnaires.
* Subject is able to provide written informed consent prior to participation in the study.
* Diagnosed with either of the following: a) overactive bladder, or b) urinary stress incontinence.

Exclusion Criteria:

* Are currently participating or have participated within the past 30 days in any clinical investigation involving or impacting urinary or renal function.
* Subject has demonstrated or is believed to be at risk of non-compliance with study procedures (e.g., for completing the diary or returning for required follow-up visits).
* Subject has undergone onabotulinumtoxin-A injections of the bladder in the last twelve (12) months.
* Subject is not suitable for the study for any reason (including overall health, pre-existing conditions or medications) in the judgment of the investigator.
* Have an untreated recurrent urinary tract infection (> 2 times within the past 6 months).
* Have neurogenic disorders such as Multiple Sclerosis, ALS, or Parkinson s Disease.
* Patients with a diagnosis of painful bladder syndrome, other pelvic pain or interstitial cystitis.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-11; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Santa Cruz, Study Director — Sponsor GmbH
Locations (2):
- United States (2):
  - Skyline Urology, Sherman Oaks, California
  - Skyline Urology, Torrance, California

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 1) Stress Urinary Incontinence | 2) Overactive Bladder
Started | 6 | 10
Completed | 6 | 8
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Population: Females diagnosed with either stress urinary incontinence or overactive bladder that met the inclusion criteria
Groups:
- Total: Total of all reporting groups
Arm/Group | 1) Stress Urinary Incontinence | 2) Overactive Bladder | Total
Number analyzed (Participants) | 6 | 10 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 7 | 11
  >=65 years | 2 | 3 | 5
Sex/Gender, Customized [Number; unit: participants]
  Female | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Used the ParaPatch System With Adverse Events Through the Completion of the Study
Description: Documentation, follow-up and characterization of all adverse events in all subjects who use the ParaPatch System, through the completion of the study.
Time Frame: up to 3 weeks
Measure: Number; unit: participants
Arm/Group | 1) Stress Urinary Incontinence | 2) Overactive Bladder
Number analyzed (Participants) | 8 | 6
participants | 8 | 6

2. Secondary Outcome: Stress Incontinence Arm
Description: Percentage of participants with less daily leaks from baseline to 3 weeks.
Time Frame: up to 3 weeks
Measure: Number; unit: percentage of subjects
Arm/Group | 1) Stress Urinary Incontinence | 2) Overactive Bladder
Number analyzed (Participants) | 6 | 8
percentage of subjects | 83 | 75

3. Secondary Outcome: Overactive Bladder Arm
Description: Percentage of participants with less daily voids from baseline to 3 weeks.
Time Frame: up to 3 weeks
Measure: Number; unit: percentage of participants
Arm/Group | 1) Stress Urinary Incontinence | 2) Overactive Bladder
Number analyzed (Participants) | 6 | 8
percentage of participants | 83 | 75

ADVERSE EVENTS:
Time Frame: 3 weeks during the device usage and for 1 week after completing device usage
Arm/Group | 1) Stress Urinary Incontinence | 2) Overactive Bladder
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No